CLINICAL TRIAL: NCT05802693
Title: An Open Clinical Study to Evaluate the Safety, Tolerance and Initial Efficacy of Epidermal Growth Factor Receptor Variant III Chimeric Antigen Receptor T(EGFRvIII CAR-T) in the Treatment of Recurrent Glioblastoma
Brief Title: A Study to Evaluate the Safety, Tolerance and Initial Efficacy of EGFRvIII CAR-T on Glioblastoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Beijing DCTY Biotech Co.,Ltd. (Other)
Responsible Party: Principal Investigator, Xuejun Yang, Chief physician, Beijing Tsinghua Chang Gung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A03728
Record Dates: First submitted 2023-03-16; First posted 2023-04-06 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The dose increase phase of this study adopts a 3+3 half-step design (Experimental): The main research objective of active comparator is to observe the efficacy and safety of Epidermal Growth Factor Receptor Variant III Chimeric antigen receptor T cells(EGFRvIII CAR-T cells) injected by local administration (Omaya capsule administration) in the treatment of Glioblastoma(GBM).
  Initial dose 22 × 10^6 cells will adopt accelerated titration (ATD); 60 × 10^6 cells，160 × 10^6 cells and 220 × 10^6 cells will use the BOIN method to increase the dose. The planned dose increase scheme is divided into accelerated titration stage (ATD) and BOIN stage
  Interventions: Drug: Targeted Epidermal Growth Factor Receptor Variant III(EGFRvIII) autochimeric antigen receptor T cell injection

INTERVENTIONS:
Drug: Targeted Epidermal Growth Factor Receptor Variant III(EGFRvIII) autochimeric antigen receptor T cell injection — Infusion of Epidermal Growth Factor Receptor Variant III Chimeric antigen receptor T(EGFRvIII CAR-T) with Omaya capsule
  Other Names: DCTY0801 Autologous T lymphocyte injection

SUMMARY:
This is a single-center, open, dose-increasing study. For subjects with recurrent glioblastomaIt ,is estimated that about 22 subjects will be enrolled, The main purpose was to evaluate the safety and tolerance of Epidermal Growth Factor Receptor Variant III Chimeric antigen receptor T(EGFRvIII CAR-T) in the treatment of patients with recurrent glioblastoma.The secondary purpose is to preliminarily evaluate the anti-tumor activity of Epidermal Growth Factor Receptor Variant III Chimeric antigen receptor T(EGFRvIII CAR-T) in the treatment of patients with recurrent glioblastoma, and preliminarily evaluate the relationship between the clinical efficacy, safety and pharmacokinetics of Epidermal Growth Factor Receptor Variant III Chimeric antigen receptor T cells(EGFRvIII CAR-T cells) preparation, as well as their correlation with tumor markers or other potential biomarkers.

This clinical study is an open clinical study, including dose increasing stage and expansion stage. The main objective of the study was to observe the efficacy and safety of Epidermal Growth Factor Receptor Variant III Chimeric antigen receptor T cells(EGFRvIII CAR-T cells) in the treatment of Glioblastoma (GBM) by local administration (Omaya capsule administration). The study will be divided into the following stages: screening stage, baseline stage, treatment stage, short-term follow-up and long-term follow-up stage.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 70 years old, gender unlimited;
2. Patients with recurrent glioblastoma confirmed by histology or cytology after surgery and treated with STUPP regimen (TMZ concurrent radiochemotherapy and adjuvant chemotherapy regimen);
3. According to the response assessment in neuro-oncology(RANO) standard, tumor lesions with evaluable or measurable (measurable enhancement lesions are defined as enhancement lesions with clear boundary on CT or MRI, which can be developed on ≥ 2 axial films with a thickness of 5 mm, and the length and diameter of each other are more than 10 mm. If the scanning layer thickness is large, the minimum measurable lesion should be more than 2 times the layer thickness);
4. Clinical pathology (immunohistochemical staining) confirmed the positive expression of EGFRvIII in the tumor;
5. Sufficient peripheral blood can be obtained through vein, and there is no other contraindication for lymphocyte collection; The peripheral blood cells can be collected according to the requirements of cell preparation;
6. KPS score ≥ 70 points;
7. Estimated survival time ≥ 3 months;
8. Subjects must give informed consent to the test before the test, and the written informed consent form shall be signed voluntarily by themselves (or their legal representatives).-

Exclusion Criteria:

1. Those who have received radiotherapy after recurrence;
2. They received immunosuppressive or glucocorticoid treatment within 2 weeks before enrollment;
3. Those who receive live vaccine within 4 weeks before enrollment and/or plan to participate in the trial;
4. He received other chemical drugs except lymphocyte clearance within 2 weeks before enrollment;
5. Not recovered from the adverse events caused by previous anti-tumor treatment before enrollment (according to NCI-CTCAE v5.0, recovered to ≤ 1 level), excluding hair loss and sequelae;
6. Previously received targeted drug therapy, cell therapy, gene therapy or other immunotherapy;
7. Have received organ transplantation in the past;
8. Those who are unable to perform brain MRI examination;
9. Any of the following exceptions occurred in the laboratory inspection:

   1. Blood routine test: absolute neutrophil count (ANC) < 1.5 × 10 ⁹/L, or platelet (PLT) < 80 × 10 ⁹/L, or hemoglobin (HGB) < 100 g/L;
   2. Coagulation function: prothrombin time (PT), or activated partial thromboplastin time (APTT), or INR > 1.5 × ULN；
   3. Liver function: total bilirubin (TBIL)>2 × ULN (upper limit of normal value), or alanine transferase (ALT), aspartate transferase (AST) > 3 × ULN；
   4. Renal function: serum creatinine (Cr) ≥ 1.5 × ULN, or glomerular filtration rate (GFR) < 60ml/min · 1.73m2;
   5. Subjects with active hepatitis B after treatment (HBsAg positive and HBV-DNA more than 1000 copies/ml (200 IU/ml) or higher than the lower detection limit, whichever is higher) are required to receive anti hepatitis B virus treatment during the study treatment; Active hepatitis C subjects (HCV antibody positive and HCV-RNA level higher than the lower limit of detection), human immunodeficiency virus or acquired immunodeficiency syndrome (HIV) related diseases. Note: Hepatocellular carcinoma(HCC) subjects with Hepatitis B virus(HBV) may be included in the study only after the researchers determine that their hepatitis is in a clinical stable state; No HCC subjects undergoing treatment are allowed to be enrolled with HCV;
   6. Cardiac ultrasound: left ventricular ejection fraction Left ventricular ejection fraction(LVEF)<50%;
10. Acute bacterial or fungal infection requiring intravenous antibiotics during cell transfusion;
11. Negligent compensatory heart failure (NYHA grade III and IV), unstable angina pectoris, acute myocardial infarction, persistent and clinically significant arrhythmia occurred within 3 months before enrollment;
12. Those who need to inhale oxygen to maintain blood oxygen saturation above 95% before entering the group and cannot return to normal within 2 weeks;
13. Having other malignant tumors and not being effectively controlled;
14. Have a history of tuberculosis;
15. Those who are known or expected to have allergic reactions or have a history of allergy to any component of the test treatment;
16. Known contrast agent allergy;
17. Have a clear history of mental disorders in the past;
18. Previous history of drug abuse or drug abuse;
19. Pregnant or lactating women, or those who plan to become pregnant during the study period;
20. Women of childbearing age and men with fertility cannot take effective and adequate contraceptive measures (such as intrauterine devices, condoms, spermicidal gel plus condoms, diaphragms, etc.) during the period of receiving the study drug and three months after the end of the study;
21. Those who participated in other clinical trials within 30 days before study enrollment;
22. The investigator judged that it was not suitable to participate in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 15 years
  Will assess dose limiting toxicity and all toxicities. Toxicity is the primary endpoint and will be assessed using the National Cancer Institute (NCI)'s Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 . Rates and associated 95% Clopper and Pearson binomial confidence limits (95% confidence interval [CI]) will be estimated for participants' experiencing dose limiting toxicity (DLT). All toxicities and side effects will be summarized in tables by dose, time period, organ, and severity.
Dose-limiting toxicity (DLT) | Up to 28 days
  A toxicity that causes side effects that are serious enough to prevent an increase in dose or level of that treatment.

SECONDARY OUTCOMES:
T cell levels | Up to 15 years
  Will assess chimeric antigen receptor (CAR) T levels and phenotype detected in peripheral blood (PB) (absolute number per ul by flow).
  Will assess EGFRvIII CAR gene copies in peripheral blood (PB)（Q-PCR method ). Statistical and graphical methods will be used to describe persistence and expansion.
Cytokine levels in PB | Up to 15 years
  Statistical and graphical methods will be used to describe persistence and expansion.
Disease response | Up to 15 years
  By Response Assessment in Neuro-Oncology (RANO) criteria with the need for Avastin as an additional indicator of progression.
Time to progression | Up to 15 years
  Progression is defined by RANO with the need for Avastin as an additional indicator of progression.
Complete response (CR) | Up to 15 years
  Kaplan Meier methods will be used to estimate median CR and graph the results.
Partial Response (PR) | Up to 15 years
  Kaplan Meier methods will be used to estimate median PR and graph the results.
Stable disease (SD) | Up to 15 years
  Kaplan Meier methods will be used to estimate median SD and graph the results.
Progressive disease (PD) | Up to 15 years
  Kaplan Meier methods will be used to estimate median PD and graph the results.
Progression free survival (PFS) | Up to 15 years
  Kaplan Meier methods will be used to estimate median PFS and graph the results.
Overall survival (OS) | Up to 15 years
  Kaplan Meier methods will be used to estimate median OS and graph the results.
Quality of life (QOL) | Up to 15 years
  Will estimate the mean and standard error for change from baseline during treatment and post treatment in the quality of life functioning scale, symptom scale and item scores from the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30（EORTC QLQ-C30）. Health-Related Quality of Life and Sympotoms will be assessed from the International Validation Study of the EORTC Brain Cancer Module(EORTC QLQ-BN20)

IPD SHARING:
Plan to Share IPD: No